CLINICAL TRIAL: NCT02319317
Title: Promoting Teen Health: A Web-based Intervention to Prevent Risky Driving
Brief Title: Web-based Intervention to Prevent Risky Driving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R00NR013548 (NIH); R00NR013548 (NIH); 14-011336 (Other: Children's Hospital of Philadelphia IRB); 821064 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2014-12-08; First posted 2014-12-18 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Adolescent; Accidents, Traffic; Attention; Motor Vehicles

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risky driving prevention (Experimental): Web-based behavioral intervention to promote teen driver attention to the roadway, addressing mobile technology and passengers.
  Interventions: Behavioral: Risky driving prevention
- Control group (Experimental): Web-based behavioral intervention for healthy lifestyles.
  Interventions: Behavioral: Control group general health promotion

INTERVENTIONS:
Behavioral: Risky driving prevention — The web-based intervention to prevent risky driving targets knowledge, attitudes, perceived control and norms about driver inattention, with strategies to keep attention on the roadway.
  Arms: Risky driving prevention
Behavioral: Control group general health promotion — The control group will receive a web-based intervention for general health promotion and is designed to enhance participants' knowledge and ability to reduce their risk of adverse health conditions including, obesity and heart disease.
  Arms: Control group

SUMMARY:
The specific aim of this study is to assess the feasibility of a web-based intervention to prevent risky driving with teen drivers licensed in the previous 90 days.

DETAILED DESCRIPTION:
The specific aim of this study is to assess the feasibility of a web-based intervention to prevent risky driving teen drivers licensed in the previous 90 days. The intervention will focus on promoting teen driver attention to the roadway.

The investigators will use a randomized controlled trial (RCT) experimental design for this feasibility study, randomizing to the intervention or control group. The investigators will complete a baseline assessment and follow up with participants at 1-month, 3-months and 6-months post-intervention delivery.

This study will provide information on the feasibility of the web-based intervention to prevent risky driving and estimation of effect size of the intervention on simulated driving performance, self-reported driving behaviors, crash and citation data.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 16-17 years at time of enrollment (i.e. can turn 18 while enrolled in research and still be eligible).
2. Pennsylvania driver's license for 90 days or less at time of assent
3. Personal email address and computer and internet access
4. Willingness to travel to CHOP twice to complete simulated assessment
5. Ability to read and write English

Exclusion Criteria:

1. Self-reported of claustrophobia, migraine headaches, or motion sickness
2. Self-reported current pregnancy
3. . Participation in a Center for Injury Research and Prevention teen driving study with the past 6 months

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine C McDonald, PhD, RN, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] McDonald CC, Sommers MS, Fargo JD, Seacrist T, Power T. Simulated Driving Performance, Self-Reported Driving Behaviors, and Mental Health Symptoms in Adolescent Novice Drivers. Nurs Res. 2018 May/Jun;67(3):202-211. doi: 10.1097/NNR.0000000000000270. PMID 29701615

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Confirmation of inclusion and exclusion criteria
Period: Overall Study
Arm/Group | Risky Driving Prevention | Control Group
Started | 31 | 29
Completed | 31 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risky Driving Prevention | Control Group | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 29 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.04 (0.39) | 16.92 (0.30) | 16.98 (0.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Retention of Participants
Description: Number of participants enrolled who complete Study Visit 1, Study Visit 2, Study Visit 3 and Study Visit 4.
Time Frame: Baseline (Study Visit 1) through Study Visit 4 (around 6 months).
Measure: Count of Participants; unit: Participants
Arm/Group | Risky Driving Prevention | Control Group
Number analyzed (Participants) | 31 | 29
Participants | 28 | 28

2. Secondary Outcome: Proportion of Participants Randomized
Description: Proportion of participants screened, enrolled and randomized
Time Frame: Baseline (Study Visit 1)
Reporting Status: Not Posted

3. Secondary Outcome: Adherence
Description: Adherence among the intervention and control group to the intervention.
Time Frame: Baseline (Study Visit 1) through completion of the intervention.
Reporting Status: Not Posted

4. Secondary Outcome: Simulated Driving Performance
Description: Difference between the intervention and control group on the simulated driving assessment (measures of driving performance during the simulated experimental drives).
Time Frame: Baseline (Study Visit 1) through Study Visit 3
Reporting Status: Not Posted

5. Secondary Outcome: Self-report Driving Behaviors
Description: Difference between the intervention and control group on self-report measures of driving behaviors.
Time Frame: Baseline (Study Visit 1) through Study Visit 4 (around 6 months).
Reporting Status: Not Posted

6. Secondary Outcome: Driving Citations and Crashes
Description: Difference between the intervention and control group on driving citations and crashes.
Time Frame: Baseline (Study Visit 1) through Study Visit 4 (around 6 months).
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Risky Driving Prevention | Control Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 2/31 | 0/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risky Driving Prevention (N=31) | Control Group (N=29)
Discomfort during/after driving simulation (General disorders) | 2 (2) | 0 (0) — Dizziness or Nausea during/after driving simulation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No